CLINICAL TRIAL: NCT03760042
Title: PHASE 1 RANDOMIZED, DOUBLE-BLIND, VEHICLE-CONTROLLED, INTRA-SUBJECT STUDY TO ASSESS LOCAL TOLERABILITY OF CRISABOROLE 2% OINTMENT AND VEHICLE IN HEALTHY PARTICIPANTS USING SUBJECT-REPORTED ASSESSMENTS AND OBJECTIVE MEASUREMENTS
Brief Title: Study To Assess Local Tolerability of Crisaborole 2% Ointment and Vehicle Ointment In Healthy Participants Using Subject-reported Assessments and Objective Measurements
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: C3291042
Record Dates: First submitted 2018-11-14; First posted 2018-11-30 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Using surrogate markers of skin sensitivity (current perception threshold and lactic acid stinging test responses) to stratify risk for developing application site treatment emergent adverse events (AS-TEAEs), within-subject comparisons will quantify AS-TEAE frequency and severity in healthy participants following double-blind applications of crisaborole ointment and vehicle ointment at 7 sensitive skin anatomic locations.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Crisaborole 2% ointment and matching crisaborole vehicle will be supplied by Pfizer to the CRU as packaged 60 gram tubes and labeled according to local regulatory requirements in an unblinded fashion.
  Crisaborole and vehicle ointment doses for the 14 pre-specified application sites bilaterally will be prepared by the unblinded PCRU pharmacist and provided to the blinded investigational site staff in individual dose containers. Subjects will be blinded to side of body treated with crisaborole and side of body treated with vehicle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Crisaborole RIGHT SIDE / Vehicle LEFT SIDE) (Other): Crisaborole ointment 2% applied to sensitive skin locations on right side of body. Crisaborole placebo vehicle ointment applied to sensitive skin locations on left side of body
  Interventions: Drug: Within-Subject Active vs Placebo Topical Applications
- Group B (Crisaborole LEFT SIDE / Vehicle RIGHT SIDE) (Other): Crisaborole placebo vehicle ointment applied to 7 sensitive skin sites on right side of body.
  Crisaborole ointment 2% applied to 7 sensitive skin locations on left side of body
  Interventions: Drug: Within-Subject Active vs. Placebo Topical Applications

INTERVENTIONS:
Drug: Within-Subject Active vs Placebo Topical Applications — Crisaborole 2% ointment (right side) and Placebo vehicle ointment (left side)
  Arms: Group A (Crisaborole RIGHT SIDE / Vehicle LEFT SIDE)
Drug: Within-Subject Active vs. Placebo Topical Applications — Crisaborole 2% ointment (left side) and Placebo vehicle ointment (right side)
  Arms: Group B (Crisaborole LEFT SIDE / Vehicle RIGHT SIDE)

SUMMARY:
A double-blind within-subject study to estimate observed application site adverse events following topical applications of crisaborole and vehicle in healthy participants

DETAILED DESCRIPTION:
To further understand the potential for crisaborole to evoke skin irritancy, a within-subject comparison study, C3291042 will assess the local tolerability of crisaborole 5 mg/cm² in healthy participants, who have had baseline assessments of surrogate markers of skin sensitivity-i.e. current perception threshold (CPT) measurements and standardized lactic acid stinging test (LAST) assessments. To further the clinical understanding of application site pain, responses to crisaborole ointment compared to crisaborole vehicle ointment will be assessed in comparisons based upon CPT (low versus high; symmetry versus asymmetry) and response to LAST ("stingers" versus "non-stingers"). This exploration of skin sensitivity characterizations in healthy participants exposed to crisaborole 5 mg/cm² will assess application site burning, stinging, and pain as well as other application site characteristics selected from a MedDRA-based list of terms by the participants. More advanced understanding of baseline application site sensation in healthy participants prior to higher local application rate of topical crisaborole may provide strategies for topical dermatologic product development programs striving to prevent or minimize application site sensory adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.

Exclusion Criteria:

* Prior self-reported history of any chronic relapsing inflammatory skin disease, including atopic dermatitis.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing). Any clinically significant medical conditions or history of such conditions that, in the opinion of the Investigator may place the participant at an unacceptable risk as a participant in this trial.
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* History of serious adverse reactions or hypersensitivity to any topical drug (eg, crisaborole); or known allergy to any of the test product(s) or any components (eg, lactic acid) in the test product(s) or history of hypersensitivity; or allergic reactions to any of the study preparations
* Abnormal physical findings of clinical significance or dermatological condition (eg extensive tattooing or excessive scarring at 14 sensitive skin application sites) at the Screening examination or Baseline which would interfere with the objectives of the study in the opinion of the Principal Investigator.
* Daily use of medications that could interfere with the objectives of the study (such as lidocaine, gabapentin, pregabalin, narcotics, antihistamines, oral or parenteral corticosteroids, non-narcotic analgesics and anti-inflammatories) within 1 week of screening and during the study.
* Not willing to refrain from shaving, the use of depilatories or other hair-removal activities, antiperspirants, lotions, skin creams, fragrances or perfumes, or body oils (eg, baby oil; coconut oil), use of hair products, hair gels, and hair oil in the treatment areas for 48 hours prior to admission to the PCRU and for the duration of the stay in the PCRU.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Application site treatment emergent adverse events (TEAEs) in crisaborole treated versus vehicle-treated prespecified sensitive skin sites | 3 days
  Comparison of investigator-reported (Application Site Skin Examination [0 to 3 points]) and participant-reported (Local Tolerability Assessment Scale scores [0 to 3 points]) application site TEAEs in crisaborole treated versus vehicle-treated at all 7 prespecified sensitive skin sites.

SECONDARY OUTCOMES:
Neurometric Measurement (Current Perception Threshold in mAmps) on Right-side and Left-side of Body (face, upper and lower extremities bilaterally) | 1 day
  Comparison of Current Perception Threshold (CPT) measurements in participants bilaterally (face, upper extremities, lower extremities) to summarize CPT (absolute value in milliAmperes and right-left differential in milliAmperes) prior to study drug dosing (CPT assessments performed at 5 Hz, 250 Hz, and 2000 Hz) .
Quantify Participant's response to Lactic Acid Stinging Test (LAST) utilizing the Local Tolerability Assessment Scale (ranging from 0 to 3 points) to categorize as Stinger or Non-stinger | 1 day
  Lactic Acid Stinging Test assessment showing Local Tolerability Assessment Scale score of 2 or 3 on lactic acid treated side AND a difference of at least 1 between lactic acid treated side and placebo treated side (ie, "stingers") versus Local Tolerability Assessment Scale score [ranging from 0 to 3 points] of 1 or less on lactic acid treated side (ie, "non-stingers").

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3291042&StudyName=Phase+1+Randomized%2C+Double-blind%2C+Vehicle-controlled%2C+Intra-subject+Study+To+Assess+Local+Tolerability+Of+Crisaborole+2%25+Ointment+And+Vehicle+In+Healthy+Participants+Using+Subject-reported+Assessments+And+Objective+Measurements